CLINICAL TRIAL: NCT02128373
Title: A Computer-Based Intervention for Distance Caregivers of Parents With Advanced Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3Z11; NCI-2014-00812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE3Z11; CASE 3Z11 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Stage IV Lung Cancer; Malignant Brain Tumor
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (usual care) (Active Comparator): Participants receive usual care (care from physician, physician nurse, and social worker) for 5 weeks. During the week 5 office visit, distance caregivers are not present. In the pre-physician interview patients will verbally complete the FACT, POMS-B, Tension-Anxiety subscale, Distress Thermometer. Distance caregivers will verbally complete the POMS-B, Tension-Anxiety subscale, and Distress Thermometer
  Interventions: Procedure: Usual care; Other: Distress Thermometer; Other: Profile of Mood States (POMS-B); Other: Quality of Life: Functional Assessment in Cancer Therapy - (FACT); Other: Tension-Anxiety Subscale
- Arm II (usual care with CLOSER intervention) (Experimental): Participants receive usual care (care from physician, physician nurse, and social worker) for 5 weeks. During the week 5 office visit, distance caregivers will use a computer-assisted intervention to be present electronically with video and audio feed to provide psychosocial support. In the pre-physician interview patients will verbally complete the FACT, POMS-B, Tension-Anxiety subscale, Distress Thermometer. Distance caregivers will verbally complete the POMS-B, Tension-Anxiety subscale, and Distress Thermometer. Up to 96 hours after the week 5 visit, patients and caregivers will be interviewed about their experience during the intervention
  Interventions: Procedure: Usual care; Other: computer-assisted intervention; Other: Distress Thermometer; Other: Profile of Mood States (POMS-B); Other: Quality of Life: Functional Assessment in Cancer Therapy - (FACT); Other: Tension-Anxiety Subscale

INTERVENTIONS:
Procedure: Usual care — Health care provided by physician, physician's nurse, and social worker
Other: computer-assisted intervention — Caregiver will virtually attend visit using the CLOSER intervention
  Arms: Arm II (usual care with CLOSER intervention)
Other: Distress Thermometer — Average score of a one item scale (range 0-10) where higher scores indicate more distress
Other: Profile of Mood States (POMS-B) — average score of five items scored 0-4 which describe how someone is feeling. Higher scores indicate increased discomfort
Other: Quality of Life: Functional Assessment in Cancer Therapy - (FACT) — Average score of FACT which quantitatively assesses brain cancer patient's physiological functional and quality of life. FACT questions are scored 0-4 with higher numbers indicating more functionality
Other: Tension-Anxiety Subscale — six item scale which asks to qualitatively describe which areas in you life are causing stress

SUMMARY:
This pilot clinical trial studies the feasibility and effectiveness of a new computer-based communication intervention in supporting distance caregivers of patients with advanced lung or brain cancer. Unlike local caregivers, distance caregivers often receive little, if any, professional support and have limited communication with the oncology team. Using a computer-based communication intervention to allow distance caregivers the opportunity to participate in a physician visit, have questions and concerns addressed, and meet members of the oncology team may help reduce stress.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. What is the relationship of primary stressors (type and stage/grade of cancer, and patient quality of life [QOL]) and structural factors/stressors (age, gender, race, and education) with patient and caregiver psychological outcomes at baseline? II. What are the effects of the Communication with Long Distance Caregivers Offering a Supportive Electronic Resource (CLOSER) intervention on distance caregiver psychological outcomes (anxiety and distress), controlling for primary stressors (type and stage/grade of cancer, and patient quality of life), distance caregiver structural factors/stressors (caregiver age, gender, race, and employment), and baseline anxiety and distress? III. What are the effects of the CLOSER intervention on patient psychological outcomes (anxiety and distress), controlling for primary stressors (type and stage/grade of cancer, and patient quality of life), distance caregiver structural factors/stressors (caregiver age, gender, race, and employment), and baseline anxiety and distress? IV. What is the feasibility (time, cost, resources and acceptability to patients, caregivers and clinicians) of using Adobe Connect, a computer-based web communication system, with the distance caregiver, the parent with advanced cancer, and the health care providers together in a routine follow-up oncology office visit? V. What is the experience of being a distance caregiver participating in the CLOSER intervention?

OUTLINE: Participants are assigned to 1 of 2 arms.

ARM I: Participants receive usual care for 5 weeks. During the week 5 office visit, distance caregivers are not present.

ARM II: Participants receive usual care for 5 weeks. During the week 5 visit, distance caregivers virtually attend using the CLOSER intervention with computer video and audio connection.

After completion of study, participants are followed up within 48-96 hours.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR PATIENTS:

* Having a diagnosis of advanced lung cancer or malignant brain tumor for two to six months
* Receiving on-going care from the medical oncologist at the Seidman Cancer Center
* Having a primary and distance caregiver involved in their care, support, and/or care planning
* English as a primary language
* Capacity to provide informed consent, as validated by the oncologist

INCLUSION CRITERIA FOR DISTANCE CAREGIVERS:

* Family caregiver of a patient with advanced lung cancer or malignant brain tumor
* Patient and distance caregiver perception that this caregiver's geographic location is such that precludes routine participation in medical appointments
* English as primary language
* Capable of providing informed consent
* Computer ownership with internet access

Exclusion Criteria:

EXCLUSION CRITERIA FOR PATIENTS:

* No primary caregiver
* Enrolled in hospice

EXCLUSION CRITERIA FOR DISTANCE CAREGIVERS:

* Those who routinely participate in most of the patient's medical appointments (once or more per month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary stressors (type and stage/grade of cancer, and patient QOL) | Baseline
  Regression analysis will be run to explore the influence of primary stressors and structural factors on patient and caregiver outcomes (anxiety and distress).
effect of CLOSER intervention on caregiver anxiety | Up to 96 hours after week 5 visit
  A two sample t-test will be conducted to compare differences in baseline to post-treatment POMS-B scores between the usual care and intervention caregiver groups
Frequency of technological errors | Up to 96 hours after week 5 visit
  Will be used to determine the feasibility of using Adobe's computer-based web communication system.
Length of time of physician office visit | Up to 96 hours after week 5 visit
  Will be used to determine the feasibility of using Adobe's computer-based web communication system.
Perceived ease of use | Up to 96 hours after week 5 visit
  Will be used to determine the feasibility of using Adobe's computer-based web communication system.
effect of CLOSER intervention on caregiver distress | Up to 96 hours after week 5 visit
  A two sample t-test will be conducted to compare differences in baseline to post-treatment Distress Thermometer scores between the usual care and intervention caregiver groups
effect of CLOSER intervention on patient distress | Up to 96 hours after week 5 visit
  A two sample t-test will be conducted to compare differences in baseline to post-treatment Distress Thermometer scores between the usual care and intervention patient groups
effect of CLOSER intervention on patient anxiety | Up to 96 hours after week 5 visit
  A two sample t-test will be conducted to compare differences in baseline to post-treatment POMS-B scores between the usual care and intervention patient groups

CONTACTS AND LOCATIONS:
Overall Officials: Sara Douglas, RN, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States